CLINICAL TRIAL: NCT06968754
Title: The Impact of Pharmaceutical Care on the Infection Control Measures Among Hemodialytic Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sulaimani (Other)
Responsible Party: Principal Investigator, Kawa Ahmad Obeid, Assistant professor, University of Sulaimani
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PH 140-24
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Infection; Hemodialysis Patients
Keywords: Pharmaceutical Care; Infection; hemodialysis; Staphylococcus aureus
MeSH Terms: conditions — Infections; Staphylococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-Intervention group (No Intervention)
- Intervention Group (Experimental): Pharmaceutical care will be provided by a clinical pharmacist in addition to conventional care. This includes assessment and resolution of drug therapy problems (DTPs) related to indication, effectiveness, safety, and compliance. Infection control interventions involve: patient education for early AV fistula use, topical antimicrobials at the catheter exit site (e.g., Mupirocin), antiseptic/antibiotic lock solutions to prevent bloodstream infections, and antimicrobial selection based on culture sensitivity. Patients will receive ongoing follow-up and support throughout the study period.
  Interventions: Other: Intervention Group

INTERVENTIONS:
Other: Intervention Group — Pharmaceutical care will be provided by a clinical pharmacist in addition to conventional care. This includes assessment and resolution of drug therapy problems (DTPs) related to indication, effectiveness, safety, and compliance. Infection control interventions involve: patient education for early AV fistula use, topical antimicrobials at the catheter exit site (e.g., Mupirocin), antiseptic/antibiotic lock solutions to prevent bloodstream infections, and antimicrobial selection based on culture sensitivity. Patients will receive ongoing follow-up and support throughout the study period.
  Arms: Intervention Group

SUMMARY:
The study aims to assess the effectiveness of pharmaceutical care in reducing infection rates among hemodialysis patients with central venous (CV) lines. It will evaluate the role of clinical pharmacists in optimizing infection management and antimicrobial use. Additionally, the study will examine the impact of pharmacist-led education on patient adherence to infection prevention and medication regimens. The role of pharmacists in reducing catheter-related bloodstream infections (CRBSIs) and other dialysis-related infections will also be investigated. Finally, the study will evaluate patient satisfaction and quality of life improvements resulting from pharmaceutical interventions in infection management.

DETAILED DESCRIPTION:
This interventional randomized controlled trial aims to investigate the impact of clinical pharmacist intervention on infection control measures among hemodialysis patients. A total of 70 patients will be randomly assigned to either an intervention group (35 patients) or a non-intervention (control) group (35 patients), and the study will be conducted over a period of six months. Patients in the intervention group will receive pharmaceutical care in addition to standard care, with the clinical pharmacist identifying and resolving drug therapy problems (DTPs) related to indication, effectiveness, safety, and compliance. Specific infection control strategies in this group will include early referral to a nephrologist and patient education to reduce catheter use, thereby promoting timely transition to permanent vascular access options such as arteriovenous fistulas or grafts. In addition, topical antimicrobial ointments (e.g., Polysporin triple antibiotic ointment, Mupirocin, or medicinal honey) will be recommended for application at the catheter exit site during insertion and at each dialysis session to reduce catheter-related bloodstream infections. Antiseptic lock solutions will be used to prevent catheter colonization and biofilm formation, while prophylactic antibiotic-anticoagulant lock solutions will be applied to further reduce bloodstream infection risk. The pharmacist will also ensure appropriate selection and monitoring of antimicrobial agents based on culture sensitivity results. Meanwhile, patients in the non-intervention group will receive only conventional healthcare, with the researcher following them regularly to assess infection rates and identify any DTPs without intervening. For both groups, regular monitoring will include laboratory tests such as CBC, C-reactive protein (CRP) plasma viscosity, blood culture, and serum creatinine.

ELIGIBILITY:
Inclusion Criteria:

* Patients in dialysis center with CKD
* Patients that can communicate with the researcher.

Exclusion Criteria:

* The patients who are not willing to participate in this study are going to be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Infection Parameters | From enrollment to about 6 months
  This study measures several clinical outcomes related to catheter use in hemodialysis patients. The primary outcome is the rate of catheter-related infections, identified based on clinical symptoms (such as fever or local inflammation) and confirmed by laboratory culture.

SECONDARY OUTCOMES:
Hospital admission rate | From enrollment to about 6 months
  Secondary outcomes include the hospital admission rate for any cause, ICU admission rate due to clinical deterioration (particularly from catheter-related sepsis), and the total length of hospital stay in days, including both ward and ICU durations. Additionally, all-cause mortality is recorded, capturing deaths from infection, dialysis-related complications, or other comorbidities. Data for all outcomes are obtained from hospital medical records and, when necessary, national death registries. These measures provide a comprehensive view of the clinical impact of the intervention and are used to compare the intervention and non-intervention groups over the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Shar Hospital, Sulaymaniyah, Sulaymaniyah Governorate, Iraq

IPD SHARING:
Plan to Share IPD: Undecided